CLINICAL TRIAL: NCT02572869
Title: Functional and Aesthetic Outcomes After Mandible Reconstruction With Fibula Osteomyocutaneous Free Flaps
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-244
Record Dates: First submitted 2015-10-01; First posted 2015-10-09 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Head and Neck Cancer
Keywords: Mandible Reconstruction; Fibula Osteomyocutaneous Free Flaps; Quality of Life; 15-244
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Restraint, Physical; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- segmental mandibulectomy and free fibular flap reconstruction: Patients who underwent segmental mandibulectomy and free fibular flap reconstruction at MSK between 1987 and 2014
  Interventions: Other: physical exam; Behavioral: questionnaires

INTERVENTIONS:
Other: physical exam — Patients will be examined by the treating physician or his/her designee (Fellow). The examining physician will complete an 11-item clinical examination form about the patient's clinical function. This examination assesses lip competence, tongue movement, oral mucosa, dental state, mouth opening, speech, drooling, diet, appearance, oral sensation, and shoulder movement. Where appropriate, the physician will ask the patient questions regarding items on the questionnaire to ensure the completeness and accuracy of the outcome assessment.
Behavioral: questionnaires — The participating patients will be asked to complete three questionnaires:
  (1) The European Organization for Research and Treatment of Cancer (EORTC) Head and Neck questionnaire (EORTC H&N 35) to assess their quality of life as it relates to their mandible function and aesthetic appearance (2) The EORTC QLQ-C30, which assesses overall health-related quality of life (3) The FACE-Q Oncology Module: Mandibulectomy, which contains questions regarding both functional and aesthetic outcomes.

SUMMARY:
The purpose of this study is to assess the functional and esthetic outcomes in patients who had removal of a part of the lower jaw bone due to mouth cancer and reconstruction of the jaw bone with a bone ( fibula) from the leg at MSKCC between the years 1987 to 2014.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write in the English language
* Patients who underwent segmental mandibulectomy and free fibular flap reconstruction at MSK between 1987 and 2014
* Able to travel to the MSK outpatient clinic or have access to email, the MSK patient portal and a computer with a camera for the follow up examination by a physician and completion of the questionnaires.

Exclusion Criteria:

* Patients who underwent marginal mandibulectomy
* Patients who underwent mandibular reconstruction with a different type of vascularized bone free flap
* Patients who underwent mandibular reconstruction with soft tissue free flap

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients will be identified from the institutional databases. Preliminary queries indicate that approximately 61 patients are eligible and currently alive.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Long-term functional (11-item clinical examination form which documents the patient's oral function) | 1 year
  The examining physician will then complete an 11-item clinical examination form which documents the patient's oral function. This examination assesses lip competence, tongue movement, oral mucosa, dental state, mouth opening, speech,drooling, diet, appearance, oral sensation, and shoulder movement.
Long-term aesthetic outcome evaluated by photographs | 1 year
  archival patient photographs taken shortly after the reconstructive surgery will be compared with photographs taken at the time of study assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jatin Shah, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/